CLINICAL TRIAL: NCT06084325
Title: The Role of Oxytocin and Interoception in Functional Neurological Disorder
Status: Completed | Type: Observational
Sponsor: University of Fribourg (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-00469
Record Dates: First submitted 2023-09-20; First posted 2023-10-16 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Functional Neurological Disorder
MeSH Terms: conditions — Conversion Disorder | interventions — Electrocardiography; Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 7.5 ml of blood (2 x 3.4ml EDTA) are taken from the test persons. The DNA is then extracted from the blood using the QIAamp DNA Blood Mini Kit (QIAGEN, Germany).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- FND Patients: Group of patients with functional neurological disorders
  Interventions: Device: Respiration resistance sensitivity task (RRST); Behavioral: Heartbeat Tracking (HBT); Device: Heartbeat evoked potential (HEP); Device: Libet task
- Healthy control: Age matched group control of healthy participant
  Interventions: Device: Respiration resistance sensitivity task (RRST); Behavioral: Heartbeat Tracking (HBT); Device: Heartbeat evoked potential (HEP); Device: Libet task

INTERVENTIONS:
Device: Respiration resistance sensitivity task (RRST) — The RRST measures interoception on the domain of the breath and thus allows its (non-invasive) manipulation. The RRST apparatus includes a step motor that moves a wedge piece back and forth to change the obstruction level in the breathing circuit. This fully automated apparatus will change the breathing obstruction level via a computer-controlled algorithm. The patient breath by the month though this device.
  Other Names: Respiration resistance device
Behavioral: Heartbeat Tracking (HBT) — The HBT measures interoception on the domain of the cardiovascular system, by assessing how accurate participants perceive their own heartbeat. After each time window participants will be asked how many heartbeats they counted, which will be compared to the actual heartbeat measured via electrocardiography (ECG).
  Other Names: ECG
Device: Heartbeat evoked potential (HEP) — The HEP is computed by averaging EEG signals time-locked to specific peaks of simultaneously measured ECG signals. Therefore both an ECG and an EEG will be set up for the participants. The task during the HEP is to simply focus on interoceptive tones (the own heartbeat) with a control condition of focusing on exteroceptive tones (sounds played). A further condition of HEP measurement is the cardio-audio synchronization. Hereby, participants will be instructed to passively listen to sounds presented to them via in-ear phones while further fixating the cross.
  Other Names: ECG + EEG
Device: Libet task — Additionally we also link the interoceptive domain of the breath to a well-known and established agency task measuring conscious intention. Participants will do two versions of the Libet taks while simultaneously recording their EEG and breathing signals with a respiratory belt.
  Other Names: Respiration belt + EEG

SUMMARY:
The main goal of this project is to better understand the role of oxytocin and Interoception in FND. More specifically oxytocin's association with precision weighing, prediction errors and priors in the interoceptive domains will be investigated. To this end, several methods will be employed: analysis of interoceptive accuracy and sensibility (interoceptive tasks and questionnaires), biomarkers of oxytocin (peripheral, endogenous oxytocin), genetic oxytocin markers (such as allele-frequency in the oxytonergic receptor gene), epigenetics (methylation rates of genes related to oxytocin), neuroactivity (EEG).

DETAILED DESCRIPTION:
The primary objective is to explore interoceptive processing during a behavioural (interoceptive) tasks and its association to the oxytocin (OT) system in patients affected by a functional neurological disorder (FND), in comparison to healthy controls (HC).

Concerning interoception, as primary outcome, it is hypothesized that:

A) FND patients are less interoceptive (judged by objectively measured accuracy) compared to HC in the interoceptive tasks.

Concerning OT, as primary outcome, it is hypothesized that:

B) The OT level is correlated with interoception tasks; specifically the adaption of precision weighting

The secondary objectives are to:

* Explore the validity and reliability of different interoceptive tasks (e.g. respiratory, cardiovascular, emotional tasks)
* Explore neuronal regions associated with interoceptive processing and interoceptive accuracy in FND compared to HC
* Investigate whether FND patients have a higher interoception trait-prediction error (discrepancy between subjective and objective interoception scores) and whether this correlates with their symptom severity
* Explore the association of the breathing cycle and the voluntary initiation of mental or motor actions, and its readiness potential
* Explore peripheral biomarkers (e.g. salivary OT) in FND patients, compared to HC
* Explore the differences in (epi)genetic profile associated with the OT-system in FND compared to HC
* Investigate the association of the OT-system and traumatic childhood experience, attachment styles and sexual functioning in patients of FND compared to HC

ELIGIBILITY:
Inclusion Criteria for Patients:

* A diagnosis of FND according to DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) diagnostic criteria
* Capable of judgement
* Willing to participate in the study (by signing the informed consent form)

Inclusion Criteria for Healthy controls:

* Capable of judgement
* Willing to participate in the study (by signing the informed consent form)

Exclusion Criteria for Patients:

* Presence of comorbid disorders such as psychosis or major depression with suicidal risk
* History of actual or suspected epilepsy
* Past surgery in the brain
* Cardio-vascular disease
* Implanted Investigational Medicinal Products (e.g. cochlear implants, neurostimulators, cardiac pacemakers)
* History of alcohol or drug abuse
* For female participants: breastfeeding, pregnancy (a standard urine pregnancy test will be provided)
* <6h prior application prostaglandin
* Long QT-syndrome
* Inability to follow the procedures of the study, e.g. due to language problems

Exclusion Criteria for Healthy controls:

* History of actual or suspected epilepsy
* Past surgery in the brain
* Cardio-vascular disease
* Implanted Investigational Medicinal Products (e.g. cochlear implants, neurostimulators, cardiac pacemakers)
* History of alcohol or drug abuse
* For female participants: breastfeeding, pregnancy (a standard urine pregnancy test will be provided)
* <6h prior application prostaglandin
* Long QT-syndrome
* Inability to follow the procedures of the study, e.g. due to language problems

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: FND patients Participants who are patients will be recruited from the in- and out-patients pool of the Clinic for Neurology of the Hospital of Fribourg and the Inselspital. At both, the treating physician will identify suitable patients (i.e. patients who fulfil the clinical requirement for FND as described in the DSM-5). The treating physician will ask these patients whether they would like to be approached by the Investigator (or his/her designee) concerning a scientific study. In case of affirmative response, the Investigator will approach the patients, inform them about the study.
  Healthy control Healthy controls will be recruited among students, collaborators, and visitors of the University of Fribourg and Bern, the Hospital of Fribourg and the Inselspital. They will be recruited by flyer, by word-of-mouth and through advertisements in public media.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-01-24 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Difference of interoception behavioural scores between FND patients and Healthy controls | 1 day
  Assessment of the difference between interoception tasks scores between these groups. These scores evaluated the interoception processing abilities of patient/control.
Difference in brain electrophysiology during interoception processing between FND patients and Healthy controls | 1 day
  Assessment of the difference Evoked Related potential (ERPs) during interoception taks between these groups.
Association between oxytocin system and interoception and its difference between FND patients and Healthy controls | 1 day
  Study of the correlation between oxytocin system and interoception indices. Oxytocin system was studied with oxytocin concentration (saliva) and genetic markers (blood analysis).

SECONDARY OUTCOMES:
Oxytocin concentration (Saliva sampling) | 1 day
  During the day of the experimental session, 4 samples of saliva at different time are collected. These sample will be used to determine the concentration of oxytocin during the day (30 min post awakening, 30min after lunch, at tasks, upon the arrival for experimental session, after the completion of all tasks).
Epigenetic profile | 1 day
  Blood sample are used for genetic analysis on the oxytocin markers (such as allele-frequency in the oxytonergic receptor gene). Correlation of this with interoceptive scores.
Respiratory Resistance Sensitivity | 1 day
  Difference of accuracy between FND patients and healthy control in the respiratory resistance sensitivity task.
Behavioral measure: heartbeat counting | 1 day
  Difference of accuracy between FND patients and healthy control to count the number of their own heartbeats.
Electrophysiological measure (EEG): Heartbeat evoked potential (HEP) task1 | 1 day
  First, study the HEP difference between interoceptive tones (the own heartbeat) with a control condition of focusing on exteroceptive tones (sounds played). Then comparison between FND patients and healthy control.
Electrophysiological measure (EEG): Heartbeat evoked potential (HEP) task2 | 1 day
  First, study the difference of mismatch negativity (MMN) evoked potential either if external tone was synchronous or asynchronous with heartbeat. Then comparison between FND patients and healthy control.
Neurophysiological measures: Correlation between agency task and respiration cycle (Libet) | 1 day
  Study of the correlation between a free will key press and the state in respiration cycle. Then comparison of the results between FND patients and healthy control.
Electrophysiological measure (EEG): the readiness potential (Libet) | 1 day
  Analysing the readiness potential related with the motor movement in the implicit compared to the explicit trigger. Then comparison of the results between FND patients and healthy control.
The localization of neuronal activity derived from EEG during interoceptive tasks, and during resting state | 1 day
  Use of the EEG signal during cardiac interception task (HEP),agency task (Libet) and resting to estimate the source generator of brain activities (inverse solution).
Behavioral measure: Correlation between oxytocin and clinical questionaire | 1 day
  Correlating the scores or categories of childhood trauma, attachment style and sexual functioning to oxytocin levels.

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - Inselspital, Bern, Canton of Bern
  - University of Fribourg, Fribourg, Canton of Fribourg

IPD SHARING:
Plan to Share IPD: No